CLINICAL TRIAL: NCT06787040
Title: Beyond One Option for the Treatment of Severe Traumatic Brain Injury [BOOTStraP]: A Pilot Study
Brief Title: Beyond One Option for the Treatment of Severe Traumatic Brain Injury
Acronym: BOOTStraP
Status: Completed | Type: Observational
Sponsor: Meditech Foundation (Other)
Collaborators: NIHR Global Health Research Group on Neurotrauma (Unknown); Gates Cambridge (Other)
Responsible Party: Principal Investigator, Andres M. Rubiano, Principal Investigator, Meditech Foundation
Other Study IDs: U1111-1272-0282
Record Dates: First submitted 2022-01-26; First posted 2025-01-22 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Traumatic Brain Injury
Keywords: TBI; LMIC; Colombia; Resource-Stratified Guidelines
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Before Implementation: Patients managed before the implementation of the stratified protocol for TBI care in the Emergency Room, Surgery, and ICU
- After Implementation: Patients managed after the implementation of the stratified protocol for TBI care in the Emergency Room, Surgery, and ICU
  Interventions: Other: Resource-Stratified Protocol

INTERVENTIONS:
Other: Resource-Stratified Protocol — The interventions are a set of protocols that accounts for varying levels of resources available at any given time for patients with severe traumatic brain injury across prehospital, ED, neurosurgery, and ICU. Protocols are available in the NIH-PMC website at: https://pmc.ncbi.nlm.nih.gov/articles/PMC7055642/
  Groups: After Implementation

SUMMARY:
Severe traumatic brain injury (sTBI) is a public health issue with great disparity among low- and middle-income countries where the implementation of evidence-based guidelines is challenging because resources are often unavailable. A consensus process including experts in the prehospital, emergency department, neurosurgery, and intensive care unit took place in Colombia to develop a set of stratified protocols called BOOTStraP, targeting resource-poor environments, but it has not been systematically implemented and tested. To identify the facilitators of, and barriers to, collecting data about patients with sTBI and to implement a stratified protocol across the treatment phases of prehospital, emergency department, neurosurgery, and intensive care unit in low-resource settings. We also aim to identify a possible association between adherence to these protocols and outcomes for these patients. A prospective, observational, before and after, pilot study will be performed in three phases as follows: before implementation, implementation, and after implementation. The BOOTStraP protocols will be implemented in three Colombian centers. We expect to find numerous barriers during the implementation phase. We also expect moderate adherence to the protocols. However, we expect to find an increase in the survival rate to hospital discharge and an improvement in neurological outcomes at discharge. This pilot study will serve as a first step to identify variables that are critical to successful implementation, to be considered for the design of a future large-scale international study to measure the effectiveness of resource-based protocols and to improve outcomes from sTBI.

DETAILED DESCRIPTION:
While evidence-based guidelines for the management of sTBI exist, their applicability in low-resource environments is limited, as the resources required to follow guidelines are often unavailable. To address this gap, a consensus process involving clinical experts was conducted in Colombia to develop a series of management protocols to articulate treatment options for TBI specific to different levels of resources and complexity across the prehospital, emergency department (ED), neurosurgery and intensive care (ICU) phases. The set of protocols was called BOOTStraP [Beyond One Option for Treatment of Traumatic Brain Injury: A Stratified Protocol]. The BOOTStraP protocols are divided into four main categories, which are based on 13 recommendations from 20 clinical experts as follows: 1) management in a basic or advanced ambulance (pre-hospital setting), 2) ED care in a low or medium-high complexity institution with or without access to a CT-Scan, 3) neurosurgery department, and 4) intermediate or ICU availability. Each one is subcategorized according to the TBI severity and can be used as a guiding tool by health professionals (e.g. EMS technicians, nurses, physicians, etc.) The user can select from a menu of treatment options depending upon resource availability (medicine, equipment, clinician training, and skill) to follow best practices given the prevailing circumstances.

This is a prospective, observational, before and after study, pilot investigation of the treatment process and outcomes for patients with TBI, who are transported by any means to a medical center for treatment. Data will be collected for each patient through the four phases of prehospital, ED, neurosurgery, and ICU, or until the patient expires. Data will be abstracted from hospital medical records.

From the initiation of the "before" phase, data for each patient will be collected from the initial patient encounter to hospital discharge, for 3 months. The BOOTStraP protocol will be implemented during the month following the end of initial data collection. After implementation ("after" phase), data for each patient will be collected from initial patient encounters to hospital discharge, for 3 months. The treatment protocols to be implemented at each center are available in the open-access published paper at the NIH PMC website: (https://pmc.ncbi.nlm.nih.gov/articles/PMC7055642/).

Each day during active data collection, the Data Collector (DC) for each site arrives at the hospital, accesses the ED records, and identifies patients admitted during the previous 24 hours who may meet inclusion criteria for the study. The DC ascertains information about the potential included patients from ED records and attending caregivers, and identifies those screened and excluded, and those screened and included. Data are transcribed from ED records and caregiver interactions directly into a web-based database. The DC completes data abstraction for included patients. The DC identifies the location and status of newly included patients, and transcribes data about each patient into the database, up to and including the current status. After completing data abstraction for new patients entered within the previous 24 hours, the DC identifies the location and status of patients previously included in the study, and transcribes data about each patient into the database, up to and including the current status. Each day during active data collection, the Study Coordinator (SC) accesses the electronic records and reviews new data entries for errors and missing data. Twice monthly, the SC visits each study site, compares abstracted data with chart records, and meets with the site DC to discuss errors and missing data. The SC and DC make any revisions together, directly into the database. During these visits, the SC records narrative information about reasons for errors and missing data, what is working and not working, and the DCs' perspectives on the barriers to and facilitators of conducting the study. The SC transcribes this narrative information into a qualitative data collection/analysis database. Categorical data will be summarized as frequencies and percentages, while continuous variables will be summarized using mean, median, minimum, maximum, and 25th and 75th percentiles. We will record narrative information from personnel at each site to investigate the barriers to and facilitators of data collection and intervention implementation. These data will be entered into a qualitative data analysis instrument, and Grounded Theory will be utilized to identify common themes. Adherence will be derived by tracking if each recommended BOOTStraP resource was available (yes/no), and if yes, whether it was utilized (yes/no). The analysis of adherence will be presented by treatment phase (prehospital, emergency department, neurosurgery, and intensive care unit). The percentage of adherence to the BOOTStrap protocol will be used as a summary statistic. The study is descriptive in nature and outcome data will be summarized descriptively by phase (before and after). The analysis will explore correlations between adherence levels by phase and individual treatments on outcome data. No hypothesis will be tested. The sample size for the study was determined based on feasibility and no formal calculation of power was performed. Implementation of BOOTStraP should increase survival to hospital discharge, and improve GOS-E at discharge. We expect there will be many barriers to implementation, especially in the pre-hospital stage. We expect adherence to protocols to be modest. This study will provide the basis to plan for a larger multi-center international study.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 15 years of age
* Clinical indications of TBI
* GCS ≤ 8 on hospital arrival, or within 48 hours of admission OR GCS ≥9 on hospital arrival, but who are either admitted to the ICU or undergo surgery within 48 hours of admission

Exclusion Criteria:

* Patient is expired at scene on EMS arrival (patients who expire during transport, either by EMS or private means, are included)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with TBI in Colombia
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Survival to hospital discharge | From date of injury until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  Evaluation of survival and mortality
Glasgow Outcome Scale Extended at discharge | From date of injury until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  Evaluation of the GOSE from 1 to 8, with 1 as the worst outcome and 8 as the best outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Andres M Rubiano, MD, Study Director — Meditech Foundation; Peter J Hutchinson, MD, PhD, Study Director — University of Cambridge
Locations (3):
- Colombia (3):
  - Clinica Uros Neiva, Neiva, Huila Department
  - Clinica Putumayo, Puerto Asís, Putumayo Department
  - Clinica La Sagrada Familia, Armenia, Quindío Department

IPD SHARING:
Plan to Share IPD: Yes
Full data of the study will be available upon request to the main contacts.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 01-01-2024 to 01-01-2029
Access Criteria: Protocol available at: https://pubmed.ncbi.nlm.nih.gov/35485862/
URL: http://www.meditechfoundationglobal.org

REFERENCES:
- [Background] Rubiano AM, Vera DS, Montenegro JH, Carney N, Clavijo A, Carreno JN, Gutierrez O, Mejia J, Ciro JD, Barrios ND, Soto AR, Tejada PA, Zerpa MC, Gomez A, Navarrete N, Echeverry O, Umana M, Restrepo CM, Castillo JL, Sanabria OA, Bravo MP, Gomez CM, Godoy DA, Orjuela GD, Arias AA, Echeverri RA, Paranos J. Recommendations of the Colombian Consensus Committee for the Management of Traumatic Brain Injury in Prehospital, Emergency Department, Surgery, and Intensive Care (Beyond One Option for Treatment of Traumatic Brain Injury: A Stratified Protocol [BOOTStraP]). J Neurosci Rural Pract. 2020 Jan;11(1):7-22. doi: 10.1055/s-0040-1701370. Epub 2020 Mar 3. PMID 32140001
- [Background] Griswold DP, Carney N, Ballarini NM, Fernandez LL, Kolias A, Hutchinson PJ, Rubiano AM. Protocol for a Multicenter, Prospective, Observational Pilot Study on the Implementation of Resource-Stratified Algorithms for the Treatment of Severe Traumatic Brain Injury Across Four Treatment Phases: Prehospital, Emergency Department, Neurosurgery, and Intensive Care Unit. Neurosurgery. 2022 Aug 1;91(2):355-359. doi: 10.1227/neu.0000000000002004. Epub 2022 May 3. PMID 35485862
- [Background] Jayaraman S, Ozgediz D, Miyamoto J, Caldwell N, Lipnick MS, Mijumbi C, Mabweijano J, Hsia R, Dicker R. Disparities in injury mortality between Uganda and the United States: comparative analysis of a neglected disease. World J Surg. 2011 Mar;35(3):505-11. doi: 10.1007/s00268-010-0871-z. PMID 21181159
- [Background] Rubiano AM, Carney N, Chesnut R, Puyana JC. Global neurotrauma research challenges and opportunities. Nature. 2015 Nov 19;527(7578):S193-7. doi: 10.1038/nature16035. PMID 26580327
- [Background] Passmore JW, Nguyen LH, Nguyen NP, Olive JM. The formulation and implementation of a national helmet law: a case study from Viet Nam. Bull World Health Organ. 2010 Oct 1;88(10):783-7. doi: 10.2471/BLT.09.071662. Epub 2010 Aug 30. PMID 20931064
- [Background] Global Status Report on Road Safety 2018: Summary. World Health Organization; 2018:20.
- [Background] Alarcon JD, Gich Saladich I, Vallejo Cuellar L, Rios Gallardo AM, Montalvo Arce C, Bonfill Cosp X. [Mortality in Colombia traffic accidents. Comparative study with other countries]. Rev Esp Salud Publica. 2018 Jul 5;92:e201807040. Spanish. PMID 29967318
- [Background] Liu BC, Ivers R, Norton R, Boufous S, Blows S, Lo SK. Helmets for preventing injury in motorcycle riders. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD004333. doi: 10.1002/14651858.CD004333.pub3. PMID 18254047
- [Background] Association WM. Declaration of Helsinki. Accessed November 26, 2021. https://www.wma.net/ policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research- involving-human-subjects/